CLINICAL TRIAL: NCT05979610
Title: Reiki-Brachy: An Interventional Treatment Trial Using Reiki Therapy to Improve Symptoms Associated With Brachytherapy in Patients With Gynecological Malignancies
Brief Title: Using Reiki Therapy to Improve Symptoms Associated With Brachytherapy in Patients With Gynecological Malignancies
Acronym: Reiki-Brachy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI158391
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Gynecologic Neoplasm; Brachytherapy; Therapeutic Touch; Endometrial Cancer; Cervical Cancer; Vaginal Cancer; Vulvar Cancer
Keywords: Reiki
MeSH Terms: conditions — Genital Neoplasms, Female; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Subjects who meet all criteria for enrollment will be randomly assigned to receive Reiki therapy (Arm 1) or usual care (Arm 2) using block randomization. Subjects will be randomized through the OnCore system in a 1:1 ratio to Arm 1 or Arm 2 and stratified by treatment type (multichannel vaginal cylinder (MCVC) and vaginal cylinder vs. all other treatment modalities). Randomization will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki Therapy (Experimental): Participants randomized to Arm 1 will receive a session of Reiki therapy during the standard wait time between the placement of the brachytherapy device and their first brachytherapy treatment.
  Interventions: Other: Reiki therapy
- Standard of Care (No Intervention): Participants randomized to the standard of care control arm will be asked to remain in a clinic room during the standard waiting period between the placement of the brachytherapy device and the start of brachytherapy treatment. Participants may participate in any activity other than Reiki therapy during this time. Participants may be accompanied by a family member or friend.

INTERVENTIONS:
Other: Reiki therapy — Reiki therapy is a form of energy healing that originated in Japan. It involves the transfer of energy from the Reiki practitioner to the recipient through the hands, with the goal of promoting physical, emotional, and spiritual well-being. Below is a general outline of the process of Reiki therapy, which may vary slightly depending on the needs of the recipient:
  * The patient will be in a quiet clinic room lying in the supine position with calming music playing and aromatherapy if the patient chooses.
  * The Reiki therapist will place their hands on or near the recipient's body. The Reiki therapist may use a series of hand positions that correspond to different energy centers in the body.
  * During the treatment, the practitioner channels energy into the recipient's body through their hands. The patient may feel a sense of warmth, tingling, or relaxation.
  * The Reiki therapist may use different techniques, such as hand movements or visualization.
  Arms: Reiki Therapy

SUMMARY:
The goal of this open label, randomized, controlled clinical trial is to assess the benefits of providing Reiki therapy to subjects receiving their first brachytherapy treatment for gynecological malignancies.

Participants will either receive a session of Reiki therapy or usual care during the standard wait time between the placement of the brachytherapy device and brachytherapy treatment. Questionnaires will be administered at various time points on the day of the participant's first brachytherapy treatment as well as at the three month follow-up time point.

Researchers will compare the intervention (Reiki therapy) and control (usual care) groups to assess the impact of the Reiki therapy on anxiety, pain, state anxiety, depression, and physiological measurements.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥ 18 years.
* Pathologically confirmed malignancy of the endometrium, cervix, vagina or vulva.
* Eligible to undergo brachytherapy treatment as an outpatient procedure.
* Able to read and understand English and/or Spanish.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Willing to participate in either the Reiki therapy or standard of care arm regardless of treatment assignment.

Exclusion Criteria:

* Prior brachytherapy treatment for a gynecological malignancy.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between the treatment groups of the change in anxiety from Assessment 1 to Assessment 3 as measured by the 6-item Spielberger State Anxiety Scale. | 4 months
  To assess the impact of Reiki therapy on anxiety in subjects undergoing brachytherapy treatment for gynecological malignancies compared to the usual care control arm.
  The 6-item Spielberger State Anxiety Scale is a validated shortened version of the Spielberger State-Trait Anxiety Inventory (STAI) used to measure state anxiety. The scale utilizes a Likert scale with four response categories assigned numerical values from 1-4 ("not at all,""somewhat,""moderately," and "very much").

SECONDARY OUTCOMES:
Comparison between the treatment groups of the change in pain from Assessment 1 to Assessment 3 as measured by the Visual Analog Scale - Pain. | 4 months
  To assess the impact of Reiki therapy on pain in subjects undergoing brachytherapy treatment for gynecological malignancies compared to the usual care control arm.
  The Visual Analogue Scale (VAS) uses an 11-point scale ranging from 0 (no symptom) to 10 (worst possible symptom). Using the pain-VAS scoring system, 0 is considered no pain, 1 - 3 is considered mild, 4 - 6 is moderate to severe, 7 - 9 is very severe and 10 is categorized as worst possible pain.
Comparison between the treatment groups of the change in anxiety from Assessment 2 to Assessment 3 as measured by the 6-item Spielberger State Anxiety Scale. | 4 months
  To assess the impact of Reiki therapy on pain in subjects undergoing brachytherapy treatment for gynecological malignancies compared to the usual care control arm.
  The 6-item Spielberger State Anxiety Scale is a validated shortened version of the Spielberger State-Trait Anxiety Inventory (STAI) used to measure state anxiety. The scale utilizes a Likert scale with four response categories assigned numerical values from 1-4 ("not at all,""somewhat,""moderately," and "very much").
Comparison between the treatment groups of the change in anxiety from Assessment 1 to Assessment 3 as measured by the Visual Analog Scale - Pain. | 4 months
  To assess the impact of Reiki therapy on pain in subjects undergoing brachytherapy treatment for gynecological malignancies compared to the usual care control arm.
  The Visual Analogue Scale (VAS) uses an 11-point scale ranging from 0 (no symptom) to 10 (worst possible symptom). Using the pain-VAS scoring system, 0 is considered no pain, 1 - 3 is considered mild, 4 - 6 is moderate to severe, 7 - 9 is very severe and 10 is categorized as worst possible pain.
Comparison between the treatment groups of the change in state anxiety and depression from Assessment 1 to three month post-radiation as measured by the Hospital Anxiety and Depression Scale. | 4 months
  To assess the impact of Reiki therapy on state anxiety and depression in subjects undergoing brachytherapy treatment for gynecological malignancies compared to the usual care control arm.
  The Hospital Anxiety and Depression Scale (HADS) is a validated, self-assessment instrument used to identify caseness of anxiety disorders and depression in medical patients. It is comprised of 14 total questions, each of which are rated on a 4-point severity scale between zero (no impairment) and three (severe impairment). Total score range is 0 (normal/no impairment) to 21 (abnormal/severe impairment.)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Burt, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No